CLINICAL TRIAL: NCT04469335
Title: Comparative Clinical Trial With Double-blind Randomized Sham Control and Additive Treatment Toward Efficacy of Mobile Neurofeedback for ADHD Youth : An Exploratory Study.
Brief Title: Effectiveness of a Mobile Neurofeedback for ADHD Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Childrens Hospital (Other)
Collaborators: Hanyang University (Other); Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Booog Nyung Kim, Professor, Seoul National University Childrens Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1905-145-1035
Record Dates: First submitted 2020-07-07; First posted 2020-07-14 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mobile neurofeedback (Experimental)
  Interventions: Device: mobile neurofeedback
- sham control (Sham Comparator)
  Interventions: Device: Sham mobile neurofeedback
- medication +mobile neurofeedback (Experimental)
  Interventions: Device: medication + mobile neurofeedback
- medication + sham control (Sham Comparator)
  Interventions: Device: medication + Sham mobile neurofeedback

INTERVENTIONS:
Device: mobile neurofeedback — to maximize usability and effectiveness, we would like to conduct a study that regulates theta/beta ratio using mobile app-based Neurofeedback Training Equipment (OmniCNS).
  The actual Neurofeedback training allows you to download and use the omnifit brain_Game, an application with an audio guide. After the pre-assessment, the researcher will provide guidance to subjects and carers on how to use the application, and demonstrate how to use it in practice. For 2 weeks, 4 weeks and 6 weeks, phone calls are conducted to check whether they are used or not and for any inconvenience. After 12 weeks of Neurofeedback training, the device is returned and post-evaluated.
  The application is equipped with four types of games and is instructed to use the three-day-a-week application. For Neurofeedback attention and cognitive training, use a headset with left and right frontal lobe 2 channel-EEG sensors to perform the game through feedback to see if it is concentrating well.
  Arms: mobile neurofeedback
Device: Sham mobile neurofeedback — It uses the sham devices and programs as the Neurofeedback, but it is not usually possible to obtain the expected effects of the Neurofeedback by providing random feedback regardless of actual brain waves.
  In case of Sham control group, parental education is conducted the same for each clinical evaluation, and in case of Sham control group, actual Neurofeedback is applied if patients and parents want it after the end of the study.
  Arms: sham control
Device: medication + mobile neurofeedback — The mobile needback is applied to patients who are taking methylphenidate or atomoxetine, which is a standard ADHD treatment, but have not been remissioned with more than 4 points of CGI-S.
  Arms: medication +mobile neurofeedback
Device: medication + Sham mobile neurofeedback — The sham mobile needback is applied to patients who are taking methylphenidate or atomoxetine, which is a standard ADHD treatment, but have not been remissioned with more than 4 points of CGI-S.
  Arms: medication + sham control

SUMMARY:
Objective: Verification of ADHD Treatment Effectiveness of Mobile Neurofeedback to Subjects of Child and Youth with ADHD.

Method: Mobile Neurofeedback Program is implemented for 165 ADHD patients aged 8 to 15 to verify their effectiveness by conducting pre-post evaluation. Prior to the implementation of the intervention, we conduct a survey with demographic information, behavioral characteristics, clinical global impression, neuropsychological test, brain MRI, NIRS and EEG.

The drug naive subjects are randomly assigned to the mobile Neurofeedback group or Sham control group. The subjects on medication are randomly assigned to the mobile Neurofeedback group or Sham control group, In addition to the medication being administered.

The intervention are conducted three times a week, twice a day, and 10-20 minutes for 12 weeks, and the effectiveness is assessed four times in advance, third month, sixth month and twelfth months.

However, the Sham control group were provided the same machines and programs as the Neurofeedback exercise, but feedback is generated randomly regardless of ectroencephalogram change of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* patient between the ages of 8 and 15

  * Patients diagnosed with ADHD in accordance with DSM-5 diagnostic criteria and K-SADS-PL ③ IQ 80 or higher ④ Neurofeedback or Sham treatment group include patients who have not received methylphenidate/atomoxetine medication in the past or who have been treated with methylphenidate less than a year and not taken methylphenidate/atomoxetine within four weeks of starting point of this study.

    * medication+Neurofeedback or medication+Sham treatment group include ADHD patients undergoing methylphenidate or atomoxetine medication over the past month without changes in capacity. And ADHD patients whose CGI-S scale is 4 or higher.

Exclusion Criteria:

* Patients diagnosed with congenital genetic disease

  * Patients with a clear history of acquired brain damage, such as cerebral palsy. ③ Patients with convulsions, other neurological disorders, or uncorrected sensory disorders

    * Patients with a history of schizophrenia, other childhood psychosis ⑤ IQ below 80 ⑥ Patient with obsessive compulsive disorder, major depression or bipolar disorder

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 165 (Estimated)
Dates: Start 2020-07-07 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Korean Attention Deficit Hyperactivity Disorder rating scale | baseline
Korean Attention Deficit Hyperactivity Disorder rating scale | 2nd week
Korean Attention Deficit Hyperactivity Disorder rating scale | 4th week
Korean Attention Deficit Hyperactivity Disorder rating scale | 8th week
Korean Attention Deficit Hyperactivity Disorder rating scale | third month
Korean Attention Deficit Hyperactivity Disorder rating scale | sixth month
Korean Attention Deficit Hyperactivity Disorder rating scale | twelfth month
Clinical Global Impression Scale-Severity | baseline
Clinical Global Impression Scale-Severity | 2nd week
Clinical Global Impression Scale-Severity | 4th week
Clinical Global Impression Scale-Severity | 8th week
Clinical Global Impression Scale-Severity | third month
Clinical Global Impression Scale-Severity | sixth month
Clinical Global Impression Scale-Severity | twelfth month
Children's Global Assessment Scale | baseline
Children's Global Assessment Scale | 2nd week
Children's Global Assessment Scale | 4th week
Children's Global Assessment Scale | 8th week
Children's Global Assessment Scale | third month
Children's Global Assessment Scale | sixth month
Children's Global Assessment Scale | twelfth month

SECONDARY OUTCOMES:
brain MRI | at the beginning, third month, sixth month, twelfth month
EEG power in beta band | at the beginning, third month, sixth month, twelfth month
EEG power in theta band | at the beginning, third month, sixth month, twelfth month
Near Infra-Red Spectroscopy | at the beginning, third month, sixth month, twelfth month

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Childrens' Hospital, Seoul, South Korea